CLINICAL TRIAL: NCT04112563
Title: COmparison of White Light and Linked COlor Imaging for Detection of RIght COlon Polyps: A Multi Center Prospective Randomized Tandem Colonoscopy Study
Brief Title: COmparison of White Light and Linked COlor Imaging for Detection of RIght COlon Polyps
Acronym: COCORICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, Principal investigator, Société Française d'Endoscopie Digestive
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ID-RCB 2019-A01287-50
Record Dates: First submitted 2019-09-29; First posted 2019-10-02 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Adenoma Colon; Colon Polyp; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: the patient will be randomized and included in one of two groups: WLI-LCI group: a first exploration of the right colon will be done in white light (WLI) then a second exploration will be done in LCI LCI-WLI group: a first exploration of the right colon will be done in LCI and a second exploration will be done in white light (WLI)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLI-LCI group (Active Comparator): a first exploration of the right colon will be done in white light (WLI) then a second exploration will be done in LCI
  Interventions: Procedure: exploration in white light (WLI); Procedure: Exploration in LCI
- LCI-WLI group (Active Comparator): a first exploration of the right colon will be done in LCI and a second exploration will be done in white light (WLI)
  Interventions: Procedure: exploration in white light (WLI); Procedure: Exploration in LCI

INTERVENTIONS:
Procedure: exploration in white light (WLI) — Exploration of the right colon done in white light (WLI)
Procedure: Exploration in LCI — Exploration of the right colon in linked color imaging (LCI)

SUMMARY:
Comparison of the number of adenomas missed by the first exploration of the right colon by LCI (linked color imaging) or by white light during a colonoscopy, according to the order of randomization.

DETAILED DESCRIPTION:
All patients consecutively admitted for routine colonoscopy will be included in this prospective randomized crossover study. After randomization, a first exploration of the right colon will be performed in linked color imaging (LCI) or white light imaging (WLI) depending of the randomization. Every polyp will be resected as soon it will be detected. After this first examination, colon will be explored a second time with a light system different from the one used for the first exploration. If a polyp will be detected during the second exploration, it will be counted as a polyp missed by the first exploration method.

A- Inclusion criteria:

1. Patient consecutively admitted to one of the endoscopy units for routine colonoscopy (screening, positive FIT, personal or family history of polyp or cancer, symptoms)
2. Patient whose age is greater than or equal to 18 years and less than 90 years
3. Score: ASA 1, ASA 2, ASA 3
4. No participation in another clinical study
5. Signed informed consent

Exclusion criteria:

History of recto-colic resection Inadequate preparation (none under Boston score <2) Patient referred for resection of a polyp in place, known IBD (inflammatory bowel disease) or known polyposis

B- Exclusion criteria:

1. History of recto-colonic resection
2. Inadequate preparation (none under Boston score <2)
3. Patient referred for resection of a known polyp
4. Inflammatory Bowel Disease
5. family polyposis
6. Score: ASA 4, ASA 5
7. Pregnant woman
8. Patient with coagulation abnormalities preventing polyp resection: TP <50%, Platelets <50000 / mm3, effective anticoagulation in progress, clopidogrel in progress
9. Patient unable to personally consent
10. No signed informed consent

Purposes of the study:

Compare, when exploring the number of adenomas missed by the first exploration of the right colon by LCI or by white light, according to the order of randomization.

Evaluation criteria :

Main criterion:

- Missed right colon adenomas by first exploration in LCI-WLI and WLI-LCI groups

Secondary criteria

* Rate of polyps missed by the first exploration
* Serrated polyp rate missed by the first exploration
* Advanced adenoma rate missed by the first exploration
* Comparison of ADR, SPDR, given by the first exploration technique decided by randomization

Number of patients:

The expected rate of "missed adenomas" of the colon is about 20%, based on published data. Considering as relevant an 8% reduction in this rate of "missed adenomas" of the right colon by the LCI, the expected rate for LCI is therefore 12%.

With a risk of the first species of 5% (bilateral test), a power of 80%, 329 patients per group should be included in the study. Taking into account the rate lost to follow-up of 5%, we expect a total of 700 patients.

Duration of the study:

1-2 years

ELIGIBILITY:
Inclusion Criteria:

* Patient consecutively admitted for routine colonoscopy

Exclusion Criteria:

* History of recto-colic resection
* Inadequate preparation (none under Boston score <2)
* Patient referred for resection of a known polyp
* known Inflammatory Bowel Disease (IBD) or known polyposis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
the number of missed adenomas during the first exploration of the right colon | 1 day
  Number of polyps diagnosed on the second exploration and not removed (because not diagnosed) during the first exploration

SECONDARY OUTCOMES:
The factors influencing these missed polyp rates | 1 day
  Time of exploration (in seconds)
The factors influencing these missed polyp rates | 1 day
  Boston scale (0 to 9)
The characteristics of the missed polyps | 1 day
  Size in millimeters
The characteristics of the missed polyps | 1 day
  type : Adenoma polyp / Advanced neoplasia polyp / Serrated polyp / Hyperplastic polyp
Adenoma Detection Rate (ADR) | 1 day
  given by the first exploration technique decided by randomization: percentage of colonoscopy with one or more adenoma of the right colon
Advanced Neoplasia Detection Rate (ANDR) | 1 day
  given by the first exploration technique decided by randomization: percentage of colonoscopy with one or more advanced neoplasia of the right colon
Serrated Polyp Detection Rate (SPDR) | 1 day
  given by the first exploration technique decided by randomization: percentage of colonoscopy with one or more serrated polyp of the right colon

CONTACTS AND LOCATIONS:
Overall Officials: David KARSENTI, MD, Principal Investigator — Société Française d'Endoscopie Digestive
Locations (1):
- Clinique Paris-Bercy, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No